CLINICAL TRIAL: NCT02543619
Title: Comparative Efficacy of Gow-Gates and Inferior Alveolar Nerve Block Injection Techniques on Success Rate of Anesthesia in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Efficacy of Two Injection Techniques on Success Rate of Inferior Alveolar Nerve Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AZad UMS
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Failed Mechanical Induction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gow-Gates injection (Active Comparator): An injection technique for infra alveolar nerve anesthesia
  Interventions: Other: Injection technique
- Infra alveolar nerve block injection (Active Comparator): An injection technique for infra alveolar nerve anesthesia
  Interventions: Other: Injection technique

INTERVENTIONS:
Other: Injection technique — One group received Gow-Gates technique and the other group received Infra Alveolar Nerve Block technique for their failed first one anesthesia

SUMMARY:
Forty healthy patients with including criteria who failed to infra alveolar nerve block injection (without lip numbness) have been randomly divided into two groups on a random basis and have received Gow-Gates or another inferior alveolar nerve block injection. Endodontic access cavity preparation has been initiated after complete anesthesia. If patients felt any pain during the steps of caries or dentin removal, Endodontic access cavity preparation or canal working length determination, treatment has been stopped and their pain has been measured by Heft Parker 170 mm Visual Analog Scale (Zero as no pain and 170 as maximum pain ).The data has been analyzed by Mann-U-Whitney and CHI- SQUARE tests.

DETAILED DESCRIPTION:
The aim of this study was to assess the efficacy of Gow-Gates and inferior alveolar nerve block on success rate of anesthesia in patients with irreversible pulpitis. In this prospective, randomized, double-blind study , forty healthy patients with symptomatic irreversible pulpitis and including criteria who failed to infra alveolar nerve block injection (without lip numbness) have been randomly divided into two groups on a random basis and have received Gow-Gates or another inferior alveolar nerve block injection. Their pain has been evaluated by electric pulp tester every 5 minutes for two times. Endodontic access cavity preparation has been initiated after complete anesthesia. If patients felt any pain during the steps of caries or dentin removal, Endodontic access cavity preparation or canal working length determination, treatment has been stopped and their pain has been measured by Heft Parker 170 mm Visual Analog Scale (Zero as no pain and 170 as maximum pain ). The patients have been instructed to rate any pain during each of the mentioned steps. The data have been analyzed by Mann-U-Whitney and CHI- SQUARE tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic irreversible pulpitis ( Visual Analog Scale ≥ 54) in one mandibular molar who need root canal treatment
* without systemic diseases
* non smoking
* non analgesic/sedative or any medicine consumption
* non pregnant
* non breast feeding
* the patients who received one conventional inferior alveolar nerve block and their block was failed ( without lip numbness)

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pain Score | 4 Hours
  Heft Parker 170 mm Analog Visual Scale

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Mohammadzadeh Akhlaghi, DDS, MDS, Principal Investigator — Associate Professor
Locations (1):
- Dental Branch, AZad UMS, Tehran, Tehran Province, Iran